CLINICAL TRIAL: NCT03888664
Title: Safety and Efficacy of γIFN Treatment in Friedreich Ataxia
Brief Title: Open Trail of γIFN for Friedreich Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT2015-002432-40
Record Dates: First submitted 2019-03-10; First posted 2019-03-25 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Interferon-gamma

STUDY DESIGN:
Intervention Model Description: 1st 2 weeks: gIFN 100 ugr/three times a week From the 3rd week: gIFN 200 ugr three times a week for the following 22 weeks From the 25th week: no treatment for the following 24 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FRDA patients treated with gIFN (Experimental): 1st 2 weeks: gIFN 100 ugr/three times a week From the 3rd week: gIFN 200 ugr three times a week for the following 22 weeks From the 25th week: no treatment for the following 24 weeks
  Interventions: Drug: gamma interferon

INTERVENTIONS:
Drug: gamma interferon — 1st two weeks: gIFN 100 ugr/three times a week from the 3rd week: gIFN 200 ugr/ three times a week for the following 22 weeks From the 25th week: no treatment for the following 24 weeks
  Other Names: Imukin 0.1 mg injectable solution

SUMMARY:
The investigator proposes an open label pilot study to investigate the safety and efficacy of gamma interferon (γIFN) in patients with Friedreich's Ataxia (FRDA). yIFN, an approved drug for treatment of granulomatous disease, has been shown to promote Frataxin expression in FRDA models in vitro and in vivo as well as in pilot human studies.

Safety will monitored by clinical surveillance and biohumoral periodic assessment. Efficacy will be assessed by a combination of advanced neuroimaging techniques and established clinical indicators. The investigators intend to recruit over a 6 months period 12 subject with molecularly established FRDA. The protocol builds on a recently concluded observational study which established the pattern of clinical and neuroimaging abnormalities characterizing a cohort of patients with FA. The data already acquired through such study will constitute the T-6/-12 point, and together with T0 assessment, carried out at study entrance, will provide for each patient the exact appreciation of disease actual progression over a year time. Recruited patients will receive for 6 months yIFN at a final dose of 200 ug/three times a week. Patients will be evaluated clinically after 3 and 6 months (T3 and T6) of treatment and 6 months after treatment end (T+6) and by neuroimaging at T6 and T+6. The neuroimaging protocol, based on 3 Tesla scanner, consists in functional MRI, tractography. The clinical protocol consists on specific ataxia scales administration. Regular monitoring with for eventual adverse events will be provided. Frataxin levels in the peripheral blood mononuclear cells will also be evaluated at T0, T3, T6, T+6. Furthermore, the thickness of the cardiac ventricle and retinal nerve fibre layer (RNFL) thickness with optical coherence tomography (OCT) will be performed at T0, T6, T + 6.

DETAILED DESCRIPTION:
Friedreich ataxia (FRDA) is a devastating neurodegenerative disease that affects children and young adults. Patients become progressively unable to coordinate movements and walking until severe disability ensues. Most patients develop dilated cardiomyopathy and congestive heart failure. The disease is non remissive and significantly shortens lifespan expectancy. FRDA is a genetic disease inherited in an autosomal recessive fashion. FRDA patients display abnormal GAA triplet expansions within the first intron of the frataxin gene that prevent proper gene expression. The levels of frataxin, a mitochondrial protein involved in iron metabolism and energy production, are insufficient and cells undergo prolonged stress and premature death. Mostly affected by frataxin deficiency are peripheral neurons of the dorsal root ganglia (DRG) and neurons of the cerebellar nucleus dentatus.

FRDA affects 1 in 50,000 individuals in western countries and has no approved therapy. It has recently been shown that interferon gamma (γIFN), a natural regulator of the immune response and iron metabolism, stimulates frataxin gene transcription and promotes frataxin accumulation in cells, including frataxin-defective cells derived from FRDA patients. Moreover, prolonged treatment of YG8R mice, an animal model for FRDA, with γIFN results in accumulation of frataxin in DRG neurons and significantly prevents the deterioration of the sensorimotor performances of the mice over time.

Since γIFN is also a drug available on the market as a recombinant protein (γIFN - 1b, TD Imukin® and Actimmune®), and already approved for two pediatric indications (malignant osteopetrosis and chronic granuloumatous disease), it could represent a quickly accessible therapeutic option for FRDA patients.

A major obstacle to efficiently establish efficacy of treatment in FRDA is the lack of reliable and sensitive biomarkers. Clinical indicators (disease specific scales, timed performance tests) are prone to inter-rater variability and, above all, while valid and sensitive to long term changes, they are very inefficient in capturing changes in the short time interval (months) typically used in randomized clinical trials (RCTs).

The advanced neuroimaging techniques such as Voxel-Based Morphometry (VBM), Susceptibility Weighted Imaging (SWI), Diffusion Tensor Imaging (DTI) and functional Magnetic Resonance Imaging (fMRI) could offer objective indicators of the disease progression that could serve as paraclinical end point in therapeutic trials. Surrogate end-points based on neuroimaging indicators have been extensively used in other neurological diseases such as Multiple Sclerosis, and their introduction speeded up significantly the recognition of effective treatments and their longitudinal evaluation.

In the last years, in vivo MRI studies have provided information relative to the damage of cerebellar, cerebral and spinal cord areas involved in FRDA and other genetically determined ataxias, which could be useful to monitor disease progression.

With the advent of the VBM, it is possible to quantify the degree of atrophy, to monitor it in time and to identify various pattern typical of a specific form of ataxia. Various studies have evidenced a significant correlation between the degree of the cerebellar atrophy, the severity of the clinical picture and also the duration of the disease .

A pilot study conducted in a cohort of 9 FRDA affected adolescents who underwent a 6 month treatment with deferiprone, demonstrated a significant reduction in the mean R2* signal in the cerebellar dentate nuclei, an iron tissue store index. Modifications of the fMRI pattern in response to specific tasks involving both the motor and the planning ability have also been demonstrated in FRDA patients, and fMRI based protocols could offer an adjunctive indicator of disease progression or of therapy induced modification.

Aims and purpose of the proposed investigation:

* Test safety of γIFN treatment given for 6 months at final dose of 200 mcg three times weekly in FRDA patients.
* Test the effect of γIFN treatment on disease specifc clinical scale (SARA)
* Test the effect of such treatment on a set of secondary imaging, laboratory and clinical end-points:
* fMRI changes in FRDA patients performing the finger tapping protocol

  * DTI parameters
  * Thickness of ventricular wall as measured by Ecocardiogram (EcoCG)
  * Thickness of RNFL as measured by OCT
  * Frataxin levels in cell lysates prepared from peripheral blood mononuclear cells (PBMC)
  * Changes in quality of life and disability impact measure. What previous work is this project based on? Evidence for the possible efficacy of recombinant γIFN in FRDA has been gathered both in the animal model for the disease and in FRDA patients. In FRDA patients, a recently completed Phase II trial reported significant improvement on the FARS evaluation after 3 months treatment on a 100 mcg, 3 times/weekly regimen. Moreover, another recently completed Phase II study suggests that the dosing of 200 mcg is reasonably well tolerated in FRDA patients.

An articulated MRI protocol for FRDA patients aged 12-50 which included DTI, VBM, and fMRI following a selective motor paradigm has been tested, validated and implemented in the investigators Institute. By this protocol the investigators evaluated 22 FRDA patients and 15 age and sex matched healthy controls, and found significant differences in DTI parameters (FA & MD) in the cerebellar white matter, long sensory and motor tracts, major commissural tracts, and in BOLD signal intensity and distribution of BOLD signal during performance of a finger tapping test. These latter disease specific changes were most evident in the ipsilateral cerebellar cortex. The observed changes correlated with the degree of neurological and functional impairment as measured with validated scales.

These preliminary results indicate that DTI and fMRI changes may function as efficient surrogate end-points in RCT for FRDA patients.

Design Open label pilot study. Primary safety end point: Safety of γIFN 6 month treatment at doses of 200 mcg 3 times a week Primary Efficacy end point: SARA score changes during the treatment period compared to those registered during the pre-treatment period and the post-treatment follow-up period

Secondary end-points:

o changes in: BOLD signal obtained during the selective motor task (finger tapping)

* DTI parameters (FA, MD) in the cerebellar white matter, the long and the commissural tracts
* Ventricular wall thickness (Eco CG)

  • RNFL thickness (OCT)
* Frataxin content in PBMC
* Changes in QoL measure (SF-36)
* Changes in Disability measure (WHO-DAS 2.0)

Subjects

Inclusion criteria:

* Molecularly defined FRDA,
* willingness to participate in the study and signing of the informed consent form.

In order to control for the ongoing deterioration associated with the disease, the investigators will recruit only those patients who had been already studied with the MRI protocol and the functional scales indicated below 12 months before the beginning of the present study.

Exclusion criteria:

* presence of any contraindication for MRI study,
* presence of clinically significant heart, liver or kidney disease or other medically unstable conditions.
* Known sensitivity to γIFN.
* Previous exposure to recombinant hematopoietin.
* Ongoing use of desferiprone or other specific FRDA treatmenent
* pregnancy or lactation

Study drug γIFN (Imukin 100 mcg/vial)

Treatment will be:

1. st two weeks: 100 mcg/three times a week From the 3rd week: 200 mcg three times a week for the following 22 weeks

   Imaging protocol

   The MRI examination will be administered at 4 T points:

   - T-12 to -6: for this point the data already stored along in the last year from the published invesitgators' MRI study on 18 subjects will be used

   - T0: at time of recruitment

   - T6: after 6 months of treatment

   - T+6: 6 months after treatment termination The protocol will be acquired on a 3 T scanner equipped with a 32-channel head coil and will include morphological, structural (DTI) and functional (fMRI) sequences.

   A 3D T1-weighted TFE sequence (TR/TE=8.2/3.7, voxel size= 1x1x1 mm, 150 slices) will be acquired in order to obtain morphological data suitable for volumetric analysis for voxel-based morphometry.

   The DTI data will be acquired by means of a T2-weighted EPI sequence (voxel size =2.5x2.5x2.5 mm) along 32 non-collinear directions, with multiple b-values (0, 300, 1100 sec/mm2) and will be evaluated off-line with the Tortoise dedicated software. Functional data will be acquired by means of a T2-weighted EPI sequence (TR/TE=2000/20, thickness=2.5mm, 40 slices) covering the whole brain and cerebellum.

   Functional images will be acquired during a task that implies manual coordination and precision, in order to test possible effect of the treatment over the functional organization of motor networks.

   Laboratory protocol Eco CG study will be performed at T0, T6, T+6 with established protocol. Frataxin levels monitoring will be performed at T0, T3 (after 3 months) and T6 (after 6 months).

   Clinical measures and Safety monitoring A trained neurologist will visit each patient at T0, T3, T6 and T+6 and report all vital signs and register other objective findings including adverse event (AE).

   A detailed checklist with all the known AE reported with γIFN treatment will be presented to each participant at T0, T3, T6.

   The following blood test will be performed at T0, T3, T6 :

   -Cell Blood Count, Erythrocyte Sedimentation Rate, Ca2+, Cl-, Na+, Mg2+, K+, Albumin, Globulins, Glucose, Blood Urea Nitrogen, Uric Acid, Creatinine, Aspartate Transaminase, Alanine Transaminase, Iron, Ferritin, Transferrin

   Statistical analysis For the MRI protocol, each dataset will be processed with a dedicated pipeline and appropriate software.

   The T1 volumes will be processed following the standard FMRIB Software Library (FSL) pipeline and performing VBM. As first step a study specific template of gray matter, using the routine "buildtemplateparallel" of Advanced Normalization Tools (ANTs), that performs an iterative template construction with elastic transformations will be created.

   The DTI data will be corrected for eddy currents and motion artefacts and then the diffusion tensor will be computed using the non-linear mono-exponential diffusion model, obtaining maps of "fractional anisotropy" (FA), "mean diffusivity" (MD), "radial diffusivity" (RD) and "axial diffusivity" (AD).

   To quantify the statistical differences over time, the diffusion data of all subjects will be moved to a common space through rigid, affine and diffeomorphic registrations based on the diffusion tensor itself. Using the transformations computed on the tensors, 3 different tests will be performed:

   - Tract Based Spatial Statistics (TBSS);

   - Voxel-wise statistical analysis based on permutations;

   - Statistical analysis of regions of interest (ROI) with generalized linear models (GLM).

   The fMRI data will be processed using Statistical Parametric Mapping 8 (SPM8). A first-level Fixed Effect analysis will be performed on each subject using global linear model and motion parameters as confounds. For the group-level analysis a Random Effect Analysis with contrasts obtained in the single subject step analysis will be performed. A two sample t-test will finally be computed to check differences in activations over time.

   All time-dependent data (including ROI-wise neuroimaging results) will be analyzed using multivariate linear mixed models, including timepoints as a repeated within-subject factor and included sex, age at onset, disease duration, years of education and number of GAA1 repeats within the smaller FXN allele as covariates of no interest. N case of a statistically significant (p<0.05) overall effect of time, pairwise comparisons between timepoints will be performed and corrected for multiple comparisons across pairs of timepoints. Correlation analysis will also be performed between possible modifications in SARA scores between consecutive time-points and the respective changes in the MRI derived structural and functional measures.

   References (Research Project):

   - Akhlaghi H, Yu J, Corben L, Georgiou-Karistianis N, Bradshaw JL, Storey E, Delatycki MB, Egan GF. Cognitive Deficits In Friedreich Ataxia Correlate with Micro-structural Changes in Dentatorubral Tract. Cerebellum. 2013 Oct 2.

   - Akhlaghi H, Corben L, Georgiou-Karistianis N, Bradshaw J, Delatycki MB, Storey E, Egan GF. A functional MRI study of motor dysfunction in Friedreich's ataxia. Brain Res. 2012 Aug 30;1471:138-54.

   - Boddaert N, Le Quan Sang KH, Rötig A, Leroy-Willig A, Gallet S, Brunelle F, Sidi D, Thalabard JC, Munnich A, Cabantchik ZI. Selective iron chelation in Friedreich ataxia: biologic and clinical implications. Blood. 2007 Jul 1;110(1):401-8.

   - Della Nave R, Ginestroni A, Tessa C, Salvatore E, Bartolomei I, Salvi F, Dotti MT, De Michele G, Piacentini S, Mascalchi M. Brain white matter tracts degeneration in Friedreich ataxia. An in vivo MRI study using tract-based spatial statistics and voxel-based morphometry.Neuroimage. 2008a Mar 1;40(1):19-25.

   - Della Nave R, Ginestroni A, Tessa C, Cosottini M, Giannelli M, Salvatore E, Sartucci F, De Michele G, Dotti MT, Piacentini S, Mascalchi M. Brain structural damage in spinocerebellar ataxia type 2. A voxel-based morphometry study. Mov Disord. 2008b Apr 30;23(6):899-903. doi: 10.1002/mds.21982.

   - Di Prospero NA, Baker A, Jeffries N, Fischbeck KH. Neurological effects of high-dose idebenone in patients with Friedreich's ataxia: a randomised, placebo-controlled trial. Lancet Neurol. 2007 Oct;6(10):878-86.

   - Georgiou-Karistianis N, Akhlaghi H, Corben LA, Delatycki MB, Storey E, Bradshaw JL, Egan GF. Decreased functional brain activation in Friedreich ataxia using the Simon effect task. Brain and Cognition 79 (2012) 200-208.

   - Jayakumar PN, Desai S, Pal PK, Balivada S, Ellika S, Kalladka D. Functional correlates of incoordination in patients with spinocerebellar ataxia 1: a preliminary fMRI study. J Clin Neurosci. 2008 Mar;15(3):269-77. doi: 10.1016/j.jocn.2007.06.021. Epub 2008 Jan 10.

   - Mantovan MC, Martinuzzi A, Squarzanti F, Bolla A, Silvestri I, Liessi G, Macchi C, Ruzza G, Trevisan CP, Angelini C. Exploring mental status in Friedreich's ataxia: a combined neuropsychological, behavioral and neuroimaging study. Eur J Neurol. 2006 Aug;13(8):827-35.

   - Montermini L, Richter A, Morgan K, Justice CM, Julien D, Castellotti B, Mercier J, Poirier J, Capozzoli F, Bouchard JP, Lemieux B, Mathieu J, Vanasse M, Seni MH, Graham G, Andermann F, Andermann E, Melançon SB, Keats BJ, Di Donato S, Pandolfo M (1997) Phenotypic variability in Friedreich ataxia: role of the associated GAA triplet repeat expansion. Ann Neurol 41:675-682.

   - Ormerod IE, Harding AE, Miller DH, Johnson G, MacManus D, du Boulay EP, Kendall BE, Moseley IF, McDonald WI. Magnetic resonance imaging in degenerative ataxic disorders.

   - J Neurol Neurosurg Psychiatry. 1994 Jan;57(1):51-7. Review.

   - Pfefferbaum A, Adalsteinsson E, Rohlfing T, Sullivan EV. MRI estimates of brain iron concentration in normal aging: comparison of field-dependent (FDRI) and phase (SWI) methods. Neuroimage. 2009 Aug 15;47(2):493-500.

   - Pierpaoli C, Walker L, Irfanoglu MO, Barnett A, Basser P, Chang L-C, Koay C, Pajevic S, Rohde G, Sarlls J, and Wu M. 2010, TORTOISE: an integrated software package for processing of diffusion MRI data, ISMRM 18th annual meeting, Stockholm, Sweden, #1597

   - Prakash N, Hageman N, Hua X, Toga AW, Perlman SL, Salamon N. Patterns of fractional anisotropy changes in white matter of cerebellar peduncles distinguish spinocerebellar ataxia-1 from multiple system atrophy and other ataxia syndromes. Neuroimage. 2009 Aug;47 Suppl 2:T72-81. doi: 10.1016/j.neuroimage.2009.05.013. Epub 2009 May 14.

   - Schenck JF, Zimmerman EA. High-field magnetic resonance imaging of brain iron: birth of a biomarker? NMR Biomed. 2004 Nov;17(7):433-45. Review.

   - Schmitz-Hübsch T, du Montcel ST, Baliko L, Berciano J, Boesch S, Depondt C, Giunti P, Globas C, Infante J, Kang JS, Kremer B, Mariotti C, Melegh B, Pandolfo M, Rakowicz M, Ribai P, Rola R, Schöls L, Szymanski S, van de Warrenburg BP, Dürr A, Klockgether T, Fancellu R. Scale for the assessment and rating of ataxia: development of a new clinical scale. Neurology. 2006 Jun 13;66(11):1717-20.

   - Schulz JB, Dehmer T, Schöls L, Mende H, Hardt C, Vorgerd M, Bürk K, Matson W, Dichgans J, Beal MF, Bogdanov MB. Oxidative stress in patients with Friedreich ataxia. Neurology. 2000 Dec 12;55(11):1719-21.

   - Seyer L, Greeley N, Foerster D et al. Open label study of Interferon gamma 1b (IFN-γ) in Friedreich ataxia. Acta Neurologica Scandinavica 2014 Oct 21. doi: 10.1111/ane.12337

   - Sormani MP, Bruzzi P. MRI lesions as a surrogate for relapses in multiple sclerosis: a meta-analysis of randomised trials. Lancet Neurol. 2013 Jul;12(7):669-76. doi: 10.1016/S1474-4422(13)70103-0.

   - Stankiewicz J, Panter SS, Neema M, Arora A, Batt CE, Bakshi R. Iron in chronic brain disorders: imaging and neurotherapeutic implications. Neurotherapeutics. 2007 Jul;4(3):371-86.

   - Subramony SH, May W, Lynch D, Gomez C, Fischbeck K, Hallett M, Taylor P, Wilson R, Ashizawa T; Cooperative Ataxia Group. Measuring Friedreich ataxia: Interrater reliability of a neurologic rating scale. Neurology. 2005 Apr 12;64(7):1261-2.
   * Tai G, Corben LA, Gurrin L et al. A study of up to 12 years of follow-up of Friedreich ataxia utilizing four measurement tools. JNNP 2014, Aug 11 as 10.1136/jnnp-2014-308022
   * Tomassini, B., Arcuri, G., Fortuni, S., Sandi, C., Ezzatizadeh, V., Casali, C., Condo, I., Malisan, F., Al-Mahdawi, S., Pook, M. and Testi R. (2012) Interferon gamma upregulates frataxin and corrects the functional deficits in a Friedreich ataxia model. Hum Mol Genet, 21, 2855-2861.
   * Trouillas P, Takayanagi T, Hallett M, Currier RD, Subramony SH, Wessel K, Bryer A, Diener HC, Massaquoi S, Gomez CM, Coutinho P, Ben Hamida M, Campanella G, Filla A, Schut L, Timann D, Honnorat J, Nighoghossian N, Manyam B. International Cooperative Ataxia Rating Scale for pharmacological assessment of the cerebellar syndrome. The Ataxia Neuropharmacology Committee of the World Federation of Neurology. J Neurol Sci. 1997 Feb 12;145(2):205-11.
   * Velasco-Sánchez D, Aracil A, Montero R, Mas A, Jiménez L, O'Callaghan M, Tondo M, Capdevila A, Blanch J, Artuch R, Pineda M. Combined therapy with idebenone and deferiprone in patients with Friedreich's ataxia. Cerebellum. 2011 Mar;10(1):1-8.
   * Villanueva-Haba V, Garcés-Sánchez M, Bataller L, Palau F, Vílchez J. Neuroimaging study with morphometric analysis of hereditary and idiopathic ataxia. Neurologia. 2001 Mar;16(3):105-11.
   * TORTOISE https://science.nichd.nih.gov/confluence/display/nihpd/TORTOISE

ELIGIBILITY:
Inclusion criteria:

* Molecularly defined FRDA,
* willingness to participate in the study and signing of the informed consent form.
* In order to control for the ongoing deterioration associated with the disease, the investigator will recruit only those patients who had been already studied with the MRI protocol and the functional scales indicated below approxymately 12 months before the beginning of the present study.

Exclusion Criteria:

* presence of any contraindication for MRI study,
* presence of clinically significant heart, liver or kidney disease or other medically unstable conditions.
* Known sensitivity to γIFN.
* Previous exposure to recombinant hematopoietin.
* Ongoing use of desferiprone or other specific FRDA treatments.
* Pregnancy or lactation

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06-26 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
number and severity of adverse drug reactions | 12 months
  number of AE and SAE reported by treated patients along the study. Safety of γIFN treatment given for 6 months at final dose of 200 mcg three times weekly in FRDA patients

SECONDARY OUTCOMES:
Changes in SARA score | 18 months
  changes in scores at the SARA scale assessed at various time points (from 6 moths before treatment start to 6 months after treatment stop) for each patient
change in BOLD signal obtained during the selective motor task (finger tapping) | 18 months
  intensity of BOLD signal in FRDA patients performing the finger tapping protocol at least 6 months prior to treatment start, at treatmenet start, after 6 months of treatment and 6 months after treatment discontinuation
Changes in RNFL thickness | 12 months
  Mean Thickness of RNFL and thickness in the 4 quadrants as resulting from OCT exam
Thickness of ventricular wall as measured by Ecocardiogram (EcoCG) | 12 months
  changes in ventricular and interventricular walls thickness (mm) at various time points for each patient
- Frataxin levels in cell lysates prepared from peripheral blood mononuclear cells (PBMC) | 12 monhts
  changes in Frataxin levels (intensity of frataxin band at western blot) associated with treatment
- Changes in quality of life measure. | 12 months
  scores at SF36 assessed along time in each patient
CHANGES in FA in the cerebellar white matter, the long and the commissural tracts | 18 months
  Fractional anysotropy values at selected ROI as measured at various time points in each patient
Changes in measure of disability | 12 months
  changes in WHO-DAS 2.0 scores recorede along time
Changes in Mean diffusivity (MD) in the cerebellar white matter, the long and the commissural tracts | 18 months
  MD values at selected ROI as measured at various time points in each patient

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Martinuzzi, MD, Principal Investigator — IRCCS Eugenio Medea

IPD SHARING:
Plan to Share IPD: No